CLINICAL TRIAL: NCT07250555
Title: sTudy of the bioEnergetics and fAtigue Responses of a Basketball gaMe: The TEAM Trial
Brief Title: Analysis of Bioenergetics and Fatigue Responses in Basketball (TEAM)
Acronym: TEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Southern Denmark (Other); Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: The TEAM trial
Record Dates: First submitted 2025-08-28; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Stress
Keywords: basketball; performance; blood metabolites; skeletal muscle metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BASKETBALL GROUP (Experimental)
  Interventions: Other: BASKETBALL GAME

INTERVENTIONS:
Other: BASKETBALL GAME — Participants will arrive 1.5 hours pre-game for initial vastus lateralis muscle biopsies and blood sampling under local anesthesia (20 mg/ml xylocaine without adrenalin). They will be fitted with IMU sensors and heart rate monitors. Volunteers are randomly assigned to teams(6 teams) for a full 40-minute game. During the match, physiological measurements will be performed at fixed times (pre, at half-time, and post-match) and after intense exercise periods (HR>90% max, high-speed runs>18km/h) within the four 10-min periods. Three groups provide samples: Group 1 (n=15): rest, half-time, end-game. Group 2 (n=8): rest, post-intense period in 1st/3rd periods. Group 3 (n=7): rest, post-intense period in 2nd/4th periods. Ten players serve as substitutes. Games will start at 17.00 - 18 p.m. to avoid diurnal variations and will be held under normal environmental conditions. A standardized 30-min warm-up period will be performed before each game.

SUMMARY:
The aims of the study are:

1. To examine skeletal muscle and blood metabolites during an official basketball game and to relate those to skeletal muscle performance during and after the game.
2. To investigate whether skeletal muscle and blood metabolites are related to game-induced fatigue.
3. To relate field activity during a basketball game with the responses of skeletal muscle and blood metabolites.
4. To investigate how blood lactate reflects muscle lactate concentration during a basketball game.
5. To determine whether temporary fatigue develops during a basketball game. game.

DETAILED DESCRIPTION:
The basketball players will participate in three experimental games (N = 10/game) on an indoors basketball stadium. During a 2-week familiarization period, volunteers will be familiarized with the experimental procedures and participate in very light training (at local basketball facilities) aimed at developing match tactics and team cohesion. At the end of the familiarization period and before the experimental game, participants will undergo a 3-day baseline performance testing (resting conditions) at University (Department of Physical Education and Sport Sciences, University of Thessaly) facilities. Prior to the games, the players will refrain from strenuous exercise and intake of alcohol for 48 hours and from tobacco and caffeine for 12 h. Dietary intake will be monitored with daily diet recalls for 7 days before the experimental period and will be standardized for all participants by a registered dietitian. The dietitian will also prescribe the meals and snacks on the game-day. On the day of the game, participants will arrive at the stadium 1.5 h before for resting skeletal muscle and blood sampling. For the first muscle biopsy and in preparation for later obtainment of biopsies from vastus lateralis muscle. An incision will be made under local anesthesia (20 mg/ml xylocaine without adrenalin) and covered by sterile band-aid strips and a thigh and shoulder bandages. In addition, an inertial measurement unit (IMU) and a heart rate monitor will be placed on each subject. During the match, a number of physiological measurements will be performed at fixed times (before the game, at half-time and post-match) and after intense exercise periods within the four 10-min periods of the game. Volunteers will be randomly assigned, using the sealed envelope procedure, in six teams representing all field positions and each team will play in one of three experimental games (random allocation using standard procedures) against each other in a full 40-minute game according to official regulations. A total of 10 additional players (from various playing positions) will serve as substitute players that could enter the pitch for a few minutes when a player will have to leave the court (either participate in measurements or will have completed it's pre-determined playing time or in case of an injury). Fifteen players (pre/post game measurement group) will have muscle and blood samples taken at rest, at the end of the 2nd period (half-time) and at the end of the 4th period (end of game). A second group of eight players (intense periods measurement group 1) will have muscle and blood samples collected at rest and during the first and third period of the game (immediately after an intense period of game-play). A third group of seven players (intense periods measurement group 1) will have muscle and blood samples collected at rest and during the second and fourth period of the game (immediately after an intense period of game-play). An intense exercise period of game-play is identified as a period with a heart rate of > 90% of maximal [as assessed by the maximal heart rate obtained during a graded exercise test to measure the maximal oxygen consumption (VO2max)], a high number of high-intensity runs (speed of > 18 km/h), sprints (speed of > 25 km/h) and/or jumps evaluated by a professional licensed coach. All muscle biopsies will be sampled from the vastus lateralis. All players will have their field activity and heart rate measured throughout the game using IMU units and heart rate monitors. Games will start at 17.00 - 18 p.m. to avoid diurnal variations and will be held under normal environmental conditions. A standardized 30-min warm-up period will be performed before each game. All games will be videotaped.

ELIGIBILITY:
Inclusion Criteria:

* Health status: were free of recent musculoskeletal injuries and/or illnesses (≥ 8 months before the study).
* Not consuming ergogenic supplements/medications (≥ 6 months before the study)
* Not smokers

Exclusion Criteria:

* Completion of the pre-determined participation time during the experimental game.
* Completion of all field measurements.
* Completion of all pre-determined sampling points for biological tissue.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of countermovement jump height | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using a force platform system
Bilateral strength peak force and rate of force development on mid-thigh pull | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using a dynamometer.
Measurement of maximal sprinting speed over 5 meters | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  5-m sprinting speed will be assessed on the basketball court using infrared photocells
Measurement of maximal sprinting speed over 20 meters | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  20-m sprinting speed will be assessed on the basketball court using infrared photocells
Measurement of the capacity to perform repeated sprints | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  5 x 20m repeated maximal sprints will be performed with 25 sec rest in between. Speed will be recorded using infrared photocells
Measurement of field activity variables during the basketball game | Continuous monitoring during each 40-minute game.
  Field activity will be continuously recorded during the basketball game using a microsensor inertial measurement unit (Kinexon Perform IMU).
Measurement of heart rate during the basketball game ad recording the average and maximal heart rate of the game. | Continuous monitoring during each 40-minute game.
  Field activity will be continuously recorded during the basketball game using a Team Polar Pro heart rate monitor.
Measurement of skeletal muscle glycogen content | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be assessed on muscle biopsy samples. Muscle glycogen content will be determined spectrophotometrically.
Measurement of skeletal muscle fiber-type distribution and fiber-type- specific glycogen content. | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be assessed on muscle biopsy samples by histochemical analysis
Measurement of skeletal muscle phosphocreatine levels | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be assessed on muscle biopsy samples by a flurometric assay.
Measurement of skeletal muscle lactate | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be assessed on muscle biopsy samples by a flurometric assay.
Measurement of effort and fatigue | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured by using the Borg Rating of Perceived Exertion (RPE) scale

SECONDARY OUTCOMES:
Body mass | Change from baseline (pre-game) to 40 minutes of the game
  Body mass will be measured using a beam balance
Body height | At baseline
  Body height will be measured using a beam balance with a stadiometer
Body mass index (BMI) | At baseline
  BMI will be calculated using the Quetelet's equation
Body fat (BF) | At baseline
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass (FM) | At baseline
  FM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat-free mass (FFM) | At baseline
  FFM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Bone mass density | At baseline
  Bone mass density will be measured by using Dual-emission X-ray absorptiometry
Bone mass content | At baseline
  Bone mass content will be measured by using Dual-emission X-ray absorptiometry
Dietary intake | At baseline
  Dietary intake will be assesed over a 7-day period using diet recalls
Evaluation of physical activity (PA) | At baseline
  International Physical Activity Questionnaire - IPAQ
Rest Heart Rate | At baseline
  The rest heart rate will be estimated using a heart rate monitor
Peak Maximal oxygen consumption (Peak VO2) | At baseline
  Peak VO2 will be estimated by open circuit spirometry via breath by breath method
Basketball-specific conditioning (endurance) | At baseline
  Yo-Yo intermittent endurance test 1
Basketball-specific conditioning (recovery) | At baseline
  Yo-Yo intermittent recovery test 1
Concentric and eccentric isokinetic peak torque of knee extensors and flexors of both dominant and non-dominant limbs | At baseline
  Will be measured at 60°/s using a three-repetition protocol via an isokinetic dynamometer
Maximal heart rate | Change from baseline (pre-game) to that recorded during the 40-minute game
  Will be measured using an automated online pulmonary gas exchange system via breath- by- breath analysis during a graded exercise testing on a treadmill
Measurement of blood lactate | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured in capillary blood collected from the index finger using a handheld portable analyzer
Measurement of plasma glucose concentration | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using a Clinical Chemistry Analyzer and a commercially available kit
Measurement of blood Glycerol concentration | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using a commercially available kit using a coupled enzyme assay involving glycerol kinase and glycerol phosphate oxidase, resulting in a colorimetric/fluorometric product proportional to the glycerol present.
Measurement of Plasma ammonia concentration | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be quantitatively determined on an analyzer using a commercially available kit
Measurement of Plasma potassium concentration | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using a flame photometer (Radiometer FLM3), with lithium as the internal standard
Measurement of Plasma- free fatty acid | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured spectophotometrically using an enzymatic kit
Measurement of blood hemoglobin and hematocrit | Change from baseline to the: a. 20th minute (half-time) and 40th minute (end of the game) (N=10), b. 5th minute (mid-1st period) and 25th minute (mid-3rd period) (N=10) and c. 15th minute (mid-2nd period) and 35th minute (mid-4th period) (N=10).
  Will be measured using an automated hematology analyzer
Measurement of fluid loss and intake | Change from baseline (pre-game) to 40 minutes of the game
  Will be measured using the measures of body mass (using a digital weight scale) and water consumption during a game.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Department of Physical Education and Sports Science, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No